CLINICAL TRIAL: NCT05960344
Title: Multicentre Prospective Cohort Study of Remote Lung Function Testing in Children: Validation and Comparison of Supervised and Unsupervised Spirometry
Brief Title: The SPIRO-MOTE Study
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Heather Elphick, Professor Heather Elphick, Sheffield Children's NHS Foundation Trust
Other Study IDs: SCH-2539
Record Dates: First submitted 2023-04-19; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spirometry — Supervised v unsupervised spirometry

SUMMARY:
Multicentre Prospective Cohort Study of Remote Lung Function Testing in Children: validation and comparison of supervised and unsupervised spirometry

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 5 to 16 years old
* Doctor diagnosed respiratory condition, including asthma, cystic fibrosis, PCD, bronchiectasis
* Child able to perform reliable spirometry
* Family have access to a smartphone or tablet and a second device for video consultation

Exclusion Criteria:

* Significant learning difficulties
* Other reasons for being unable to do lung function tests, for example, unable to make a seal around the mouthpiece
* Informed consent/assent has not been provided
* No English speaking member of the family
* Contraindications as outlined by the ARTP, e.g. pneumothorax, haemoptysis of unknown origin, unstable cardiovascular status, recent eye surgery, vomiting or any acute disease that would interfere with the test performance, recent surgery (thoracic/abdominal)

Ages: 5 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Participants will be recruited at the four participating centres: Sheffield Children's Hospital, Leeds Children's Hospital, Royal Hospital for Children (Glasgow) and Great Ormond Street Hospital (London).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Outcome measures from spirometry tests (1) | Within two weeks
  The researchers will use the absolute values for FEV1 and FVC, coupled with the demographic data, to calculate FEV1/FVC, percent predicted and z-scores using a batch calculator from the GLI website. The team will record how many patients achieved technically acceptable tests, using the ATS A-F standards (9), and how many failed.
Outcome measures from spirometry tests (2) | Within two weeks
  The team will record how many patients achieved technically acceptable tests, using the ATS A-F standards (9), and how many failed.
Length of each standard test | Within two weeks
  Researchers will record how long each standard test took to carry out.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No